CLINICAL TRIAL: NCT05407077
Title: Is Lower Limb Neuromotor Control Diverse in Females With PF OA Contrasted With Asymptomatic Controls When Performing Stair Descent Task?
Brief Title: Is Lower Limb Neuromotor Control Diverse in Females With PF OA Contrasted With Asymptomatic Controls
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Jilan Adel yousef, lecturer, Cairo University
Other Study IDs: P.T.REC/012/003437
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Chondromalacia Patellae
MeSH Terms: conditions — Chondromalacia Patellae

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- females with isolated patellofemoral arthritis: those with anterior knee pain
- healthy females: those without anterior knee pain

SUMMARY:
Objective: to investigate whether females with PF OA descend stairs with different muscular recruitment strategies contrasted with similar aged healthy females.

Methods: An observational comparative study will be conducted with thirty females with PF OA and 10 healthy ones. The onset times and electromyography (EMG) duration of multifidus, transversus abdominus (TrA), gluteus medius (GM), and vasti muscles will be measured by quantitative EMG during stair descent task. hypothesis: Investigators hypothesize that there won't be a significant difference between females with PF OA and their matched healthy group regarding the onset times and duration of vastus medialis obliqus (VMO), vastus lateralis (VL), gluteus medius (GM), multifidus, and transversus abdominus (TrA), during stair descent task.

DETAILED DESCRIPTION:
Investigators will collect the EMG activity of VMO, VL, GM, multifidus, and TrA using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels highresolution wireless bio amplifier (WBA) system (Biomation, Almonte, Canada). Electromyographic data will be sampled at 1000 Hz and bandpass filtered at 50-200 Hz. For each muscle, three electrodes will be used; two electrodes will be placed ~30 mm apart in the direction of the muscle fibers and a ground electrode will be placed over the closest bony prominence. Before placement of the electrodes, the subject's skin will be cleaned with alcohol to reduce impedance and excess hair will be removed to eliminate shifting of the electrodes if needed. The stair-stepping task consists of descending 2 steps. Patients should start descending the steps immediately in response to a command, at their normal speed with their affected limb. Healthy subjects should start descending stairs with their dominant limb . Before data acquisition, participants should perform one practice trial of stair descent to get familiarized with the task. Then the participants should perform three test trials with thirty seconds of rest after each trial to prevent fatigue. The raw data will be stored on a personal computer for analysis with a custom program in Matlab (Math Works, Natick, Massachusetts, USA). Investigators should use a mean of data in three trials for analysis.

ELIGIBILITY:
Inclusion Criteria:

* • Inclusion Criteria for PF OA group; patients will be included if they have

  1. Anterior- or retro-patellar knee pain aggravated by at least two activities that load the PFJ (eg; stair ambulation, squatting and/or rising from sitting) .
  2. Pain during these activities presented on most days during the past month and their pain severity was ≥ 4 on an 11 point numerical pain scale during aggravating activities .,
  3. A grade less than (2) from postero-anterior views on the Kellgren - Lawrence (KL) grading scale.

Inclusion Criteria for Healthy control subjects :

1. no history of knee pathology or pain with any of the provocative activities which were mentioned above

Exclusion Criteria:

* • Exclusion Criteria for Patients in the PF OA group:

  1. concomitant pain from tibiofemoral joint or other knee structures . • Exclusion Criteria for Subjects from both groups:

  <!-- -->

  1. current or previous pain in the hip, lumbar spine or foot that lasted longer than 3 months and/or required intervention.
  2. a history of lower extremity, pelvis or spine fractures; spine, hip, knee or foot surgeries; hip or patellar subluxation/ dislocation.
  3. injury to any of knee ligaments or meniscus.
  4. systemic diseases (e.g. rheumatoid arthritis), neurological conditions or fibromyalgia . 5.The professional athletes; people who exercise more than two hours a day or every other day.

Ages: 35 Years to 55 Years | Sex: Female
Age Groups: Adult
Study Population: Patients will be recruited from the Outpatient Clinic of Kasr Al-Ainy Hospital and the Faculty of Physical Therapy, Cairo University as well. However, control subjects will be recruited via advertising in the local community.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2023-01-02 (Actual)

PRIMARY OUTCOMES:
The change of EMG onset of multifidus | from admission to discharge, up to two weeks
  investigators will collect the EMG activity of multifidus using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels high-resolution wireless bioamplifier (WBA) system (Biomation, Almonte, Canada).
The change of EMG duration of multifidus | from admission to discharge, up to two weeks
  investigators will collect the EMG activity of multifidus using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels high-resolution wireless bioamplifier (WBA) system (Biomation, Almonte, Canada).
The change of EMG duration of transversus abdominus | from admission to discharge, up to two weeks
  investigators will collect the EMG activity of transversus abdominus using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels high-resolution wireless bioamplifier (WBA) system (Biomation, Almonte, Canada).
The change of EMG onset of transversus abdominus | from admission to discharge, up to two weeks
  investigators will collect the EMG activity of transversus abdominus using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels high-resolution wireless bioamplifier (WBA) system (Biomation, Almonte, Canada).
The change of EMG onset of gluteus medius | from admission to discharge, up to two weeks
  investigators will collect the EMG activity of gluteus medius using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels high-resolution wireless bioamplifier (WBA) system (Biomation, Almonte, Canada).
The change of EMG duration of gluteus medius | from admission to discharge, up to two weeks
  investigators will collect the EMG activity of gluteus medius using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels high-resolution wireless bioamplifier (WBA) system (Biomation, Almonte, Canada).
The change of EMG onset of vastus medialis obliqus | from admission to discharge, up to two weeks
  investigators will collect the EMG activity of vastus medialis obliqus using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels high-resolution wireless bioamplifier (WBA) system (Biomation, Almonte, Canada).
The change of EMG duration of vastus medialis obliqus | from admission to discharge, up to two weeks
  investigators will collect the EMG activity of vastus medialis obliqus using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels high-resolution wireless bioamplifier (WBA) system (Biomation, Almonte, Canada).
The change of EMG duration of vastus lateralis | from admission to discharge, up to two weeks
  investigators will collect the EMG activity of vastus lateralis using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels high-resolution wireless bioamplifier (WBA) system (Biomation, Almonte, Canada).
The change of EMG onset of vastus lateralis | from admission to discharge, up to two weeks
  investigators will collect the EMG activity of vastus lateralis using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels high-resolution wireless bioamplifier (WBA) system (Biomation, Almonte, Canada).

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy, Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No